CLINICAL TRIAL: NCT02536560
Title: "Intestinal Microbiota Composition After Antibiotic Treatment in Early Life. The INCA Study"
Brief Title: Intestinal Microbiota Composition After Antibiotic Treatment in Early Life
Acronym: INCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Agentschap NL (Other Government)
Collaborators: Danone Global Research & Innovation Center (Industry); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Nicole B.M.M. Rutten, PhD candidate, Agentschap NL
Other Study IDs: NL.37233.100.11, R-11.26AM
Record Dates: First submitted 2015-08-21; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Microbiota; Eczema; Atopy
Keywords: intestinal microbiota; antibiotics; infant; allergy
MeSH Terms: conditions — Eczema; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — faecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Antibiotics: 150 infants, (because of hospital protocol) treated with antibiotics because of a perinatal infection during the first week of life
- Controls: The control group comprises 300 healthy newborns, born in the hospital and needing clinical observation for 24-48 hours for several reasons like maternal comorbidity, low probability of neonatal infection, blood sugar monitoring, meconium containing amniotic fluid, or delivery by caesarean section

SUMMARY:
In this prospective observational cohort study the potential clinical consequences of antibiotic use in early life and perturbations in the gastrointestinal microbiota composition due to that antibiotic use are studied. It is hypothesized that altered microbiota may be an important underlying mechanism for impediments in the developing immune system.

Differentiation will be made between a group of neonates who received antibiotics in the first week of life, and control infants who were not exposed to antibiotics in the neonatal period.

DETAILED DESCRIPTION:
Healthy newborns born in the hospital, observed for low probability of neonatal infection will be compared to newborns exposed to antibiotic therapy in early life (first 1-2 weeks).

Infants are recruited from the maternity wards and neonatal wards of four teaching hospitals in the Netherlands. In total 150 infants, treated with antibiotics because of (a high suspicion of) a perinatal infection during the first week of life, will be recruited. The control group comprises 300 healthy newborns, born in the hospital and needing clinical observation for 24-48 hours for several reasons like maternal comorbidity, low probability of neonatal infection, blood sugar monitoring, meconium containing amniotic fluid, or delivery by caesarean section.

Differences in clinical outcomes between antibiotic treated infants and controls are investigated. Incidence of atopic dermatitis (eczema), food allergy, upper respiratory tract infections (URTI), lower respiratory tract infections (LRTI), gastrointestinal infections (GITI) and excessive crying are evaluated, prospectively assessed by parental reports and retrospectively assessed by doctor's diagnoses. The clinical endpoints will be linked to the developing intestinal microbiota during the first year of life.

Potential differences in intestinal fecal microbiota composition and diversity can be determined at eight time points during the first year of life, as sampling moments include: day one (T1), day two (T2), one week (T3), two weeks (T4), one month (T5), three months (T6), six months (T7), one year (T8).

ELIGIBILITY:
Inclusion Criteria:

1. Term-born babies (≥ 36 weeks gestational age)
2. (Short) stay on maternal ward or admission to neonatal ward because of antibiotic treatment
3. Signed informed consent by the parents

Exclusion Criteria:

1. Congenital illness or malformations
2. Severe perinatal infections for which transfer to the neonatal intensive care unit is needed
3. Maternal probiotic use ≤ six weeks before delivery
4. Insufficient knowledge of the Dutch language.

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy newborns born in the hospital, observed for low probability of neonatal infection will be compared to newborns exposed to antibiotic therapy in early life (first 1-2 weeks) by investigating potential differences in intestinal fecal microbiota composition
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Clinical endpoints | Participants will be followed during their first year of life
  Differences in clinical outcomes between antibiotic treated infants and controls are investigated. Incidence of atopic dermatitis (eczema), food allergy, upper respiratory tract infections (URTI), lower respiratory tract infections (LRTI), gastrointestinal infections (GITI) and excessive crying are evaluated. Data are prospectively assessed by parental reports (calendar lists).

SECONDARY OUTCOMES:
Microbiota composition | Samples will be taken at eight time points during the participant's first year of life
  Fecal bacterial composition and diversity is determined at eight time points during the first year of life, from birth on. Sampling points include: day one (T1), day two (T2), one week (T3), two weeks (T4), one month (T5), three months (T6), six months (T7), one year (T8).
  Potential differences in microbiota composition and diversity will be determined by use of 16S-23S ribosomal ribonucleic acid (rRNA) gene analysis (IS-pro).
Vaccine response | around 1 year of age
  Immunoglobulin G antibodies against Tetanus toxoid, Diphtheria toxoid, Haemophilus influenza type B, and the capsular polysaccharides of the pneumococcal 10-valent conjugate vaccine will be determined.
  Antibody concentrations will be determined from blood samples. Measured in international units per milliliter or microgram per milliliter.
Doctor's diagnosis | Participants will be followed during their first year of life
  Diagnoses are defined by selected International Classification system of Primary Care (ICPC) codes, diagnosticated during the first year of life.
  These include: dyspnea (R02), wheezing (R03), cough (R05), acute upper tract infection (R74), acute bronchi(oli)tis (R78), pneumonia (R81), asthma like symptoms (R96), breath problems [R04], sneeze [R07], other symptoms of the nose [R08], symptoms of the throat [R21], abnormal sputum [R25], concern about respiratory illness [R27], acute laryngitis [R77], influenza [R88], other infections of the airways [R83], and other respiratory diseases [R99], infectious diarrhea (D70), vomiting (D10), susceptible gastro-intestinal infection (D73), other symptoms/complaints of the skin (S21), dry skin/ flaking (S21.01), infantile colic (A14).

OTHER OUTCOMES:
infant height | Participant's height is monitored during the first year of life
  Individual height is monitored during the first year of life. Parents report the most recently measured height of the child on the calendar lists.
  (height is measured in centimeters)
infant weight | Participant's weight is monitored during the first year of life
  Individual weight is monitored during the first year of life. Parents report the most recently measured weight of the child on the calendar lists.
  (weight is measured in kilograms)
coughing | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  The child coughs several times a day and/or has coughing. Regularly there are signs of cold. Cough because of choking does not have to be recorded.
wheezing | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  During expiration the parents notice a whistling, wheezy sound coming from the lower airways of the child. During expiration the child is trying to squeeze the air outwards. Wheezing coming from or through the nose does not have to be recorded.
fever >38 degrees Celsius | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  Clear from itself, whereby it is important that parents use a rectal thermometer, measure twice and the temperature is >38 degrees Celsius on both occasions.
runny nose | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  Signs of cold with white/yellow/green mucus running from the nose.
glue ear | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  The child seems to have earache and/or grasps its ear (the ear frequently is high-colored or bends) and/or glue egresses from the ear.
rash | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  More than one day existing skin-redness (spots, rash, pimples) on the face, arms or legs, trunk. Disease-symptoms are not necessarily present. The rash can be eczema; eczema mostly is red, scaly and may itch. Infants cheeks are affected mostly. When children grow up, elbow and knees are preferred sites.
diarrhea | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  Watery or mucous defecation, more than three times a day, that continues more than one day.
>3 crying hours a day | the symptom is daily reported as present or not present (by the parents, on the calendar list), during the infant's first year of life
  Parental reported symptom on calendar list (yes/no). Description:
  Clear from itself, whereby the total crying episodes add up to more than three hours a day (24 hours) in total.
prescribed antibiotics | Participants will be followed during their first year of life and prescription of antibiotic courses will be monitored
  Any prescribed (systemic) antibiotic treatments during the first year of life are investigated. Measured as number of antibiotic courses during the first year of life, [1] parental reported (on the calendar list) and [2] checked via pharmacist's medication records.
allergic sensitization | around 1 year of age
  (serum) allergen antibodies to food and inhalant allergens are determined. Measured in kilo unit.

CONTACTS AND LOCATIONS:
Overall Officials: Arine M Vlieger, MD, PhD, Principal Investigator — St Antonius Hospital Nieuwegein, the Netherlands
Locations (4):
- Netherlands (4):
  - Gelre Hospitals, Apeldoorn, Gelderland
  - Meander Medical Centre, Amersfoort, Utrecht
  - Tergooi Hospital, Blaricum, Utrecht
  - St Antonius Hospital, Nieuwegein, Utrecht

REFERENCES:
- [Derived] Daele EV, Kamphorst K, Belzer C, van Elburg RM, Knol J, Smidt H, Vlieger AM. Aberrant microbiota signatures precede symptom development in infantile colic. J Pediatr Gastroenterol Nutr. 2025 Aug;81(2):217-225. doi: 10.1002/jpn3.70101. Epub 2025 Jun 9. PMID 40485532
- [Derived] An R, Fontana F, Van Daele E, Ventura M, Vlieger A, van Elburg RM, Knol J, Milani C, Belzer C. Longitudinal changes in bifidobacterial population during the first two years of life. Benef Microbes. 2024 Apr 30;15(3):227-240. doi: 10.1163/18762891-bja00012. PMID 38677714
- [Derived] Kamphorst K, Vlieger AM, Oosterloo BC, Garssen J, van Elburg RM. Neonatal Antibiotics and Food Allergy Are Associated With FGIDs at 4-6 Years of Age. J Pediatr Gastroenterol Nutr. 2022 Jun 1;74(6):770-775. doi: 10.1097/MPG.0000000000003428. Epub 2022 Feb 24. PMID 35588166
- [Derived] Oosterloo BC, Van't Land B, de Jager W, Rutten NB, Klopping M, Garssen J, Vlieger AM, van Elburg RM. Neonatal Antibiotic Treatment Is Associated With an Altered Circulating Immune Marker Profile at 1 Year of Age. Front Immunol. 2020 Jan 10;10:2939. doi: 10.3389/fimmu.2019.02939. eCollection 2019. PMID 31998285
- [Derived] Kamphorst K, Oosterloo BC, Vlieger AM, Rutten NB, Bunkers CM, Wit EC, van Elburg RM. Antibiotic Treatment in the First Week of Life Impacts the Growth Trajectory in the First Year of Life in Term Infants. J Pediatr Gastroenterol Nutr. 2019 Jul;69(1):131-136. doi: 10.1097/MPG.0000000000002360. PMID 31058782
- [Derived] Rutten NB, Rijkers GT, Meijssen CB, Crijns CE, Oudshoorn JH, van der Ent CK, Vlieger AM. Intestinal microbiota composition after antibiotic treatment in early life: the INCA study. BMC Pediatr. 2015 Dec 9;15:204. doi: 10.1186/s12887-015-0519-0. PMID 26645894